CLINICAL TRIAL: NCT02109081
Title: Dexamethasone and Postoperative Delirium
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Investigator left institution
Sponsor: Endeavor Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: EH13-477
Record Dates: First submitted 2014-04-05; First posted 2014-04-09 (Estimated); Last update posted 2021-12-21 (Actual); Status verified 2019-09

CONDITIONS: Delirium; Postoperative Cognitive Dysfunction
Keywords: dexamethasone; delirium; postoperative cognitive dysfunction; postoperative; elderly
MeSH Terms: conditions — Delirium; Postoperative Cognitive Complications | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexamethasone (Experimental): Patients will be administered dexamethasone 10 mg at induction of anesthesia
  Interventions: Drug: Dexamethasone
- Placebo-2.5 cc of saline (Placebo Comparator): Patients will be administed placebo at induction of anesthesia
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexamethasone
  Arms: Dexamethasone
Drug: Placebo
  Arms: Placebo-2.5 cc of saline

SUMMARY:
Postoperative delirium is commonly observed in elderly patients in the postanesthesia care unit (PACU) and during the first 2-3 days following surgical procedures. This is an important clinical problem in the geriatric surgical patient; morbidity and mortality rates are significantly higher in patients who develop delirium. At the present time, the etiology of delirium has not been precisely defined. However, studies suggest that inflammation related to the surgical stress response is an important contributing factor in inducing neuroinflammation and subsequent cognitive dysfunction and delirium. Therefore it is possible that agents which attenuate perioperative inflammation may reduce the risk of the development of delirium following surgery. Dexamethasone is a potent corticosteroid that is used by anesthesiologists primarily as an antiemetic agent. Small doses of dexamethasone have also been demonstrated to significantly reduce the release of inflammatory markers after surgery. The anti-inflammatory effects of corticosteroids have the potential to beneficially impact neuroinflammation and the risk of developing postoperative delirium. The aim of this randomized, controlled, double-blinded investigation is to determine if dexamethasone, administered at induction of anesthesia, can decrease the incidence of delirium at the time of discharge from the PACU and during the first 2 days following surgery.

DETAILED DESCRIPTION:
This study will be a randomized, placebo-controlled, double blind clinical investigation. Four hundred patients scheduled for surgical procedures under general anesthesia will be enrolled. Patients will be randomized via a computerized randomization table to one of two groups; a dexamethasone group (10 mg of dexamethasone in a 5 cc syringe) or a control group (an equal volume of saline in a 5 cc syringe)). A dose of 10 mg of dexamethasone was selected, as this reflects a dose that has been demonstrated to attenuate the inflammatory response to surgery, decrease pain, and improve clinical recovery. This is also within the dose range commonly used at NorthShore University HealthSystem. The drug/placebo solution will be prepared by the pharmacy into the syringes. Both solutions are clear and appear identical. Study syringes will be prepared by the pharmacy, and all clinicians will be blinded to group assignment. At the induction of anesthesia, the syringe containing either dexamethasone or saline will be administered. The administration of all other anesthetic agents will be standardized and reflect the usual practices of anesthesiologists at NorthShore University HealthSystem.

Monitoring will consist of standard American Society of Anesthesiologists monitors, which include manual blood pressure measurements, continuous EKG monitoring, pulse oximetry, capnography and infrared gas analysis. Additional monitoring, such as direct radial artery pressure measurements, will be at the discretion of the attending anesthesiologist. Anesthetic induction will consist of propofol 0.5-2.0 mg/kg, fentanyl 50-100 μg, and rocuronium 0.6 mg/kg. Anesthesia will be maintained with sevoflurane 0.5-3.0%, with the concentration of inhalational agent adjusted to maintain blood pressure within 20-30% of baseline values and depth of anesthesia standardized using a BIS monitor (BIS values 40-60). Additional doses of fentanyl, up to 1-2 µg/kg/hour, can be administered at the discretion of the anesthesia care provider. Hydromorphone may be provided for postoperative analgesia. Hypotension (any decrease in mean arterial pressure ≥ 20%) will be treated with a fluid bolus, phenylephrine, or ephedrine, as clinically indicated. Thirty minutes before the anticipated conclusion of the surgical procedure, patients will receive ondansetron 4 mg. Neuromuscular blockade will be reversed with neostigmine and glycopyrrolate.

Patients will be managed according to standard PACU protocols. Nausea and vomiting will be treated per standard protocols. Any episodes of nausea and vomiting in the PACU will be noted on a data collection sheet. Pain will be treated with hydromorphone. Pain scores in the PACU, as well as total doses of hydromorphone will be recorded. Patients will be discharged from the PACU when standard criteria are met. Study subjects will be discharged either to the surgical floor or the intensive care unit (ICU). The times to meet discharge criteria and actually achieve discharge will be recorded. For patients transferred directly to the ICU from the operating room, nausea, vomiting, pain scores, and analgesic requirements will be collected over the first 3 hours of recovery. Postoperatively, pain will be controlled with intravenous doses of hydromorphone. Intravenous analgesia will be provided until patients are able to resume oral intake, which usually occurs on the first or second postoperative day. At this time, analgesic management will be transitioned to oral pain medication (typically hydrocodone 5 mg / acetaminophen 500 mg). Total doses of intravenous and oral pain medications will be recorded during the hospitalization. Postoperative pain scores will be assessed at the same time testing for delirium is performed during the postoperative period. A planned interim analysis will be performed when 200 patients are enrolled

ELIGIBILITY:
Inclusion Criteria:

* patients ≥ 70 years of age, undergoing a noncardiac surgical procedure under general anesthesia, with an anticipated duration of postoperative admission of at least 2 days.

Exclusion Criteria:

* 1) preoperative diagnosis of delirium or dementia; 2) MMSE score of ≤ 20 out of 30 on preoperative testing (more than mild cognitive impairment) or delirium on preoperative CAM testing; 3) language barriers that would preclude testing; 4) preoperative steroid use within 3 days of surgery; or 5) anticipation of postoperative intubation.

Ages: 70 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2021-02 (Actual); Study Completion 2021-02 (Actual)

PRIMARY OUTCOMES:
Postoperative delirium at postanesthesia care unit (PACU) discharge | 45 minutes after PACU admission
  The Confusion Assessment Method (CAM) test will be used to determine the presence or absence of delirium. The CAM assesses the acute onset and attention deficits as primary features, and level of consciousness and disorganized thinking as secondary features. In order to measure the primary and secondary components of the CAM, additional formal testing is required; the Mini Mental State Exam (MMSE) will be used.

SECONDARY OUTCOMES:
Postoperative delirium day one | 24 hours after surgery
  The Confusion Assessment Method (CAM) test will be used to determine the presence or absence of delirium. The CAM assesses the acute onset and attention deficits as primary features, and level of consciousness and disorganized thinking as secondary features. In order to measure the primary and secondary components of the CAM, additional formal testing is required; the Mini Mental State Exam (MMSE) will be used.
Postoperative delirium day two | 48 hours after surgery
  The Confusion Assessment Method (CAM) test will be used to determine the presence or absence of delirium. The CAM assesses the acute onset and attention deficits as primary features, and level of consciousness and disorganized thinking as secondary features. In order to measure the primary and secondary components of the CAM, additional formal testing is required; the Mini Mental State Exam (MMSE) will be used.
MMSE scores at postanesthesia care unit discharge | 45 minutes after PACU admission
  The Mini Mental State Exam (MMSE) is an easy to use test of cognitive function that can be administered in 5-10 minutes. It was specifically developed to screen for dementia, with scores of ≤ 20 out of 30 indicating moderate cognitive dysfunction.
MMSE on postoperative day one | 24 hours after surgery
  The Mini Mental State Exam (MMSE) is an easy to use test of cognitive function that can be administered in 5-10 minutes. It was specifically developed to screen for dementia, with scores of ≤ 20 out of 30 indicating moderate cognitive dysfunction.
MMSE on postoperative day two | 48 hours after surgery
  The Mini Mental State Exam (MMSE) is an easy to use test of cognitive function that can be administered in 5-10 minutes. It was specifically developed to screen for dementia, with scores of ≤ 20 out of 30 indicating moderate cognitive dysfunction.
Hospital length of stay | 5 days
  The total length of the hospitalization will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Glenn S. Murphy, MD, Principal Investigator — Endeavor Health
Locations (1):
- NorthShore University HealthSystem, Evanston, Illinois, United States